CLINICAL TRIAL: NCT02333123
Title: Aspirin for Venous Ulcers: Randomised Trial (AVURT)
Acronym: AVURT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment halted following TSC meeting due to poor recruitment and study unlikely to complete. Funders withdrew continued support
Sponsor: St George's, University of London (Other)
Collaborators: University of York (Other); University of Manchester (Other); Bradford Teaching Hospitals NHS Foundation Trust (Other Government); Harrogate & District NHS Foundation Trust (Other); Hull University Teaching Hospitals NHS Trust (Other Government); University of Nottingham (Other); Cardiff University (Other); University of Newcastle Upon-Tyne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14.0096
Record Dates: First submitted 2014-11-05; First posted 2015-01-07 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Experimental): Aspirin 300mg capsule by mouth once a day for 24 weeks.
  Interventions: Drug: Aspirin
- Placebo (Placebo Comparator): Placebo capsule (for aspirin 300mg capsule) by mouth once a day for 24 weeks.
  Interventions: Drug: Placebo (for Aspirin)

INTERVENTIONS:
Drug: Aspirin — Each 300mg aspirin capsule will contain over-encapsulated 4 x Aspirin 75mg tablets.
  Arms: Aspirin
Drug: Placebo (for Aspirin) — Each placebo capsule will contain a lactose and magnesium stearate blend, and will appear identical in weight, colour and size to the matched aspirin capsules.
  Arms: Placebo

SUMMARY:
This efficacy study evaluates the safety and effectiveness of aspirin for venous leg ulcer healing. The study also examines whether patients can be recruited to a larger study. Patients with chronic venous leg ulceration presenting and undergoing care in leg ulcer community clinics or hospital out-patient clinics, or registered with a clinic but are receiving care at home will be recruited. All patients will receive standard compression bandaging. Half of the participants will be randomised to receive aspirin, while the other half will receive a placebo.

DETAILED DESCRIPTION:
The mainstay of treatment of leg ulcers is graded compression therapy to squeeze the fluid out of the leg and venous system. This has been shown to be effective in many clinical trials. However, despite this treatment patients take many months to heal (with median healing times of approximately 12 weeks in previous trials) and for some patients compression therapy does not result in resolution of their leg ulcers. The use of compression (as well as dressings largely to manage the wound exudate) can be expensive as nurse time is required to change bandages which can be required weekly or more frequently. Furthermore, for many patients the compression therapy is uncomfortable (sometimes painful) and inconvenient for everyday life (compression is bulky and dressings have to be changed several times weekly). If other treatments were able to reduce the time to healing then this would be a significant breakthrough.

Results from two earlier small trials suggest aspirin may be of benefit. However this trials were poorly designed and reported. The present study will evaluate whether the addition of 300mg of daily aspirin to standard evidence based therapies reduces the time to healing of chronic venous leg ulceration using a more rigorous design. The study will also establish the feasibility of satisfactory participant recruitment for a bigger trial, and whether participants are compliant with their aspirin therapy. The safety of aspirin in this patient population will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Those with at least one chronic venous leg ulcer - where chronic venous leg ulceration is defined as any break in the skin which has either: a) been present for more than six weeks, or b) occurred in a person with a history of venous leg ulceration. Ulcers will be considered purely venous if clinically no other etiology was suspected. For this the ulcer must be venous in appearance (i.e. moist, shallow, of an irregular shape) and lie wholly or partially within the gaiter region of the leg. If the patient has more than one ulcer we will choose the largest ulcer as the 'index' lesion for purposes of the analysis.
* Ulcer area > 1 square cm
* Participants must have had an ankle brachial pressure index (ABPI) ≥ 0.8 taken within the previous three months. When the ABPI is incompressible other forms of assessment including peripheral pulse examination / toe pressure / duplex ultrasound in combination with clinical judgement to be used to exclude PAD
* Aged ≥ 18 years (no upper age limit)
* Able and willing to provide informed consent
* Ulcer duration > 6 weeks or prior history of venous ulceration.

Exclusion Criteria:

* Unable to provide consent
* Unwilling to provide consent
* Foot (below the ankle) ulcer
* A leg ulcer of non-venous aetiology (i.e. arterial)
* Ankle-brachial pressure index (ABPI) <0.8
* Current regular use of aspirin (as may be randomised to placebo)
* Previous intolerance of aspirin / contraindication to aspirin (decision made according to the prescribers' clinical judgement)
* Prohibited medication: Probenecid
* Known lactose intolerance (as placebo contains lactose)
* Pregnant/lactating women
* Currently participating in another study evaluating leg ulcer therapies.
* Another reason that excluded them from participating within this trial (decision made according to the nurses' or prescribers' clinical judgment )*
* Previously been recruited in to this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-07-10 (Actual); Primary Completion 2016-08-18 (Actual); Study Completion 2016-11-11 (Actual)

PRIMARY OUTCOMES:
Time to healing of the reference ulcer (the largest eligible ulcer) | 25 weeks

SECONDARY OUTCOMES:
Ulcer size (area) measured in square cm | 25 weeks
Recurrence of reference ulcer | 25 weeks
  Proportion of participants with a recurrence of reference ulcer. Time to recurrence.
Ulcer related pain using the VAS Score | 5 weeks
Treatment concordance: number of participants completing the course of treatment | 24 weeks
  Proportion of participants completing the course of treatment up to healing or planned trial exit. The number of capsules taken. Nurse's assessment of participant's compliance with recommended compression therapy.
Resource use | 27 weeks
  Number and duration of all leg ulcer-related appointments with health professionals (including wound related in-patient stays ). Number of and types of dressings used.
Number of adverse events | 27 weeks
  Number of participants with at least one event. Total number of events.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Hinchliffe, MD, FRCS, Principal Investigator — St George's Healthcare NHS Trust
Locations (5):
- United Kingdom (5):
  - Hull & East Yorkshire Hospital NHS Trust, Cottingham, Castle Hill Hosp
  - St George's University Hospitals NHS Foundation Trust, Tooting, London
  - Harrogate & district NHS Trust, Harrogate, N.Yorkshire
  - Brighton General Hosp, Brighton, Sussex
  - Freeman Hospital, Newcastle upon Tyne

REFERENCES:
- [Derived] Helen T, Liz C, Laura C, Illary S, Martin B, Hannah B, Ian C, Jo D, Chris F, Rachael F, Rhian G, Keith H, Alison L, Ellie L, Catriona MD, Christine M, Debbie R, Gerard S, David T, Peter V, Laurie W, Robert H. Aspirin versus placebo for the treatment of venous leg ulcers-a phase II, pilot, randomised trial (AVURT). Trials. 2019 Jul 26;20(1):459. doi: 10.1186/s13063-019-3480-7. PMID 31349862
- [Derived] Tilbrook H, Clark L, Cook L, Bland M, Buckley H, Chetter I, Dumville J, Fenner C, Forsythe R, Gabe R, Harding K, Layton A, Lindsay E, McDaid C, Moffatt C, Rolfe D, Sbizzera I, Stansby G, Torgerson D, Vowden P, Williams L, Hinchliffe R. AVURT: aspirin versus placebo for the treatment of venous leg ulcers - a Phase II pilot randomised controlled trial. Health Technol Assess. 2018 Oct;22(55):1-138. doi: 10.3310/hta22550. PMID 30325305
- [Derived] Tilbrook H, Forsythe RO, Rolfe D, Clark L, Bland M, Buckley H, Chetter I, Cook L, Dumville J, Gabe R, Harding K, Layton A, Lindsay E, McDaid C, Moffatt C, Phillips C, Stansby G, Vowden P, Williams L, Torgerson D, Hinchliffe RJ. Aspirin for Venous Ulcers: Randomised Trial (AVURT): study protocol for a randomised controlled trial. Trials. 2015 Nov 10;16:513. doi: 10.1186/s13063-015-1039-9. PMID 26554558